CLINICAL TRIAL: NCT00057655
Title: Access to Behavioral Health Services for Women on TANF
Brief Title: Behavioral Health Services for Women Receiving Public Assistance
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R03MH065384 (NIH); R03MH065384 (NIH); DSIR SE
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Mental Disorders
Keywords: Social Welfare; Mentally Ill Persons; Mental Health Services
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether access to behavioral health services has been affected by welfare reform.

DETAILED DESCRIPTION:
This study examines patterns of behavioral health service use among a group of female household heads who receive Temporary Assistance to Needy Families (TANF) and have serious mental illness (SMI). The findings from this study will be used to determine the feasibility of conducting a full-scale longitudinal study of the impact of welfare reform outcomes on female household heads who have SMI and are currently or formerly recipients of welfare.

ELIGIBILITY:
Inclusion Criteria:

* Female head of household on TANF at any time during first quarter of 1997 and used at least one behavioral health service during that quarter
* DSM IV diagnosis of serious mental illness

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2002-01; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, School of Social Work, Philadelphia, Pennsylvania, United States